CLINICAL TRIAL: NCT05517993
Title: Effect of Gui-Lu-Er-Xian-Jiao-Wan on Intradialytic Hypotension: a Randomized Crossover Pilot Trial
Brief Title: Effect of Gui-Lu-Er-Xian-Jiao-Wan on Intradialytic Hypotension
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8M0841
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Intradialytic Hypotension
Keywords: Intradialytic Hypotension; Chinese herbal medicine; Gui-Lu-Er-Xian-Jiao

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Gui-Lu-Er-Xian-Jiao-Wan (GLEXJW) 3g orally twice daily for 12 weeks.
  Interventions: Drug: Gui-Lu-Er-Xian-Jiao-Wan
- Group B (No Intervention): No intervention.

INTERVENTIONS:
Drug: Gui-Lu-Er-Xian-Jiao-Wan — Gui-Lu-Er-Xian-Jiao-Wan (GLEXJW) is an ancient CHM formula, mainly originating from processed tortoise shells, antlers, Ginseng, and wolfberry.
  Other Names: GLEXJW
  Arms: Group A

SUMMARY:
Intradialytic hypotension (IDH), a common complication during hemodialysis (HD) could increase patients' morbidity and mortality. Previous studies considered that some Chinese herbal medicine (CHM) plays a complementary role in reducing the frequency of IDH. This trial is aimed to investigate the effect of Gui-Lu-Er-Xian-Jiao-Wan (GLEXJW) in patients with intradialytic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease treated with hemodialysis for ≥3 months
* Receive a standard thrice-weekly hemodialysis schedule
* More than 25% of hemodialysis sessions complicated by intradialytic hypotension

Exclusion Criteria:

* Active malignancy
* Life-threatening conditions
* Pregnancy
* Recent participation in another clinical trial for intradialytic hypotension
* History of hypersensitivity or contraindication to herbal medicine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Intradialytic hypotension episode | Each time of dialysis during 12-weeks study period.
  Hypotension episode during hemodialysis

SECONDARY OUTCOMES:
Early termination of hemodialysis | Each time of dialysis during 12-weeks study period.
  The episode of early termination in hemodialysis due to hypotension
SF-36 | Baseline, 12 weeks, 28 weeks
  Short Form (36) Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No